CLINICAL TRIAL: NCT05397639
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Masupirdine (SUVN-502) for the Treatment of Agitation in Participants With Dementia of the Alzheimer's Type
Brief Title: Masupirdine for the Treatment of Agitation in Dementia of the Alzheimer's Type
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP3S1502HT6; 2021-003405-22 (EudraCT Number)
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Agitation; Alzheimer's Type Dementia
Keywords: Masupirdine; SUVN-502; Phase 3; Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — 1-((2-bromophenyl)sulfonyl)-5-methoxy-3-((4-methyl-1-piperazinyl)methyl)-1H-indole dimesylate monohydrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Masupirdine Arm (Experimental): Tablet
  Interventions: Drug: Masupirdine 50 mg
- High Dose Masupirdine Arm (Experimental): Tablet
  Interventions: Drug: Masupirdine 100 mg
- Placebo (Placebo Comparator): Tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Masupirdine 50 mg — Tablet, Once Daily
  Other Names: SUVN-502
  Arms: Low Dose Masupirdine Arm
Drug: Masupirdine 100 mg — Tablet, Once Daily
  Other Names: SUVN-502
  Arms: High Dose Masupirdine Arm
Drug: Placebo — Matching Placebo Tablet, Once Daily
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the efficacy, safety, tolerability, and pharmacokinetics of masupirdine compared to placebo for the treatment of agitation in participants with dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study, consisting of 12 weeks of treatment.

Approximately 375 participants will be enrolled at approximately 50 centers worldwide.

Study medication will be administered orally once-daily from Day 1 through Day 85. Screening will occur within approximately 4 weeks prior to randomization. Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants will be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of dementia of the Alzheimer's type according to the National Institute on Aging-Alzheimer's Association (NIA-AA) criteria.
* Has confirmed agitation using the IPA Consensus Provisional Definition of Agitation in Cognitive Disorders.
* Has a score between 8 and 24 (both inclusive) on Mini-Mental State Examination (MMSE).

Exclusion Criteria:

* Participants with dementia predominantly of the non-Alzheimer's type (e.g., vascular dementia, parkinson's disease, lewy body disease, frontotemporal dementia)
* Has symptoms of agitation that are not secondary to Alzheimer's disease (eg, pain, other psychiatric disorder, or delirium due to a metabolic disorder, systemic infection, or substance-induced).
* Participant (or caregiver) is deemed otherwise ineligible for participation in this study in the investigator's judgement.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | From Baseline to Week 12 visit
  Change in CMAI items score aligning to the International Psychogeriatric Association (IPA) agitation criteria domains (physical aggression, excessive motor activity, and verbal aggression). CMAI is a validated 29-item questionnaire to assess agitation. Each item is rated on a 7-point scale ranging from 1 "Never" to 7 "Several times per hour". Higher scores indicate worsening agitation.

SECONDARY OUTCOMES:
Modified Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (mADCS-CGI-C) | From Baseline to Week 12 visit
  Change in mADCS-CGI-C. The mADCS-CGI-C is a modification of the ADCS-CGI-C instrument that focuses specifically on agitation. It is a 7-point Likert scale that ranges from marked improvement scored as 1 to marked worsening scored as 7. The range is from 1 to 7. Higher scores indicate worsening agitation.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (27):
  - Advanced Research Center, Inc., Anaheim, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Leading Edge Research LA, LLC, Encino, California
  - Neuro Pain Medical Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Mary S Easton Center for Alzheimer's Research and Care UCLA, Los Angeles, California
  - Ki Health Partners, LLC, Stamford, Connecticut
  - Allied Biomedical Research Institute, Miami, Florida
  - Central Miami Medical Institute, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Miami Jewish Health, Miami, Florida
  - Novel Clinical Research Center, LLC., Miami, Florida
  - Brainstorm Research, Miami, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Quantum Laboratories Inc, Pompano Beach, Florida
  - Re:Cognition Health, Chicago, Illinois
  - Insight Hospital and Medical Center Chicago, Chicago, Illinois
  - Ocean Medical Research, Toms River, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - Velocity Clinical Research, Cleveland, Beachwood, Ohio
  - Ralph H. Johnson VA Health Care System, Charleston, South Carolina
  - Midlands Neurology and Pain Associates, Columbia, South Carolina
  - Gadolin Research, Beaumont, Texas
  - Re:Cognition Health, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Clinical Trial Network, Houston, Texas
- Croatia (4):
  - Clinical Hospital Center Rijeka, Rijeka
  - Polyclinic Neuron, Zagreb
  - University Hospital Center Zagreb, Zagreb
  - Klinika za psihijatriju Vrapce, Zagreb
- Poland (8):
  - Medycyna Milorzab sp. z o.o., Lodz, Lódzkie
  - FutureMeds Warszawa Centrum, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research powered by Pratia, Warsaw, Masovian Voivodeship
  - Centrum Leczenia Zaburzen Pamieci Affidea, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Silmedic Sp z o o, Katowice, Silesian Voivodeship
  - EMC Silesia Sp. z o.o., Katowice, Silesian Voivodeship
  - Neuro-Medic Janusz Zbrojkiewicz, Katowice, Silesian Voivodeship
  - ClinHouse Centrum Medyczne, Zabrze
- Serbia (5):
  - Clinical Hospital Center Dragisa Misovic Dedinje, Belgrade
  - Special Hospital for Psychiatric Diseases, Kovin
  - University Clinical Center Kragujevac, Clinic for Psychiatry, Kragujevac
  - University Clinical Center Nis, Clinic for neurology, Niš
  - Clinical Centre of Vojvodina, Clinic of Neurology, Novi Sad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The study drug, Masupirdine (SUVN-502), is being investigated for the treatment of agitation associated with dementia of the Alzheimer's type. — https://agitation-study.com/